CLINICAL TRIAL: NCT03380520
Title: Effect of Intravenous FerRic carbOxymaltose oN Reverse Remodeling Following Cardiac Resynchronization Therapy
Acronym: IRON-CRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Wilfried Mullens, MD PhD, Md PhD, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRON-CRT
Record Dates: First submitted 2017-11-02; First posted 2017-12-21 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferric carboxymaltose (Experimental): Ferric carboxymaltose according to SmPC
  Interventions: Drug: Ferric Carboxymaltose
- Placebo (Placebo Comparator): Normal saline (0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric Carboxymaltose — Ferric carboxymaltose will be administered according to product specification dosing
  Other Names: injectafer
  Arms: Ferric carboxymaltose
Drug: Placebo — IV nacl 0.9%
  Arms: Placebo

SUMMARY:
To assess impact on left ventricular reverse remodeling defined as a change in left ventricular ejection fraction in heart failure patients with reduced ejection fraction (and previous implantation of cardiac resynchronization therapy) undergoing treatment with ferric carboxymaltose vs. placebo

ELIGIBILITY:
Inclusion Criteria:

1. Chronic heart failure and implantation of cardiac resynchronization therapy more than 6 months ago and presence of iron deficiency (ferritin < 100 μg/l, irrespective of TSAT or ferritine between 100 - 300 μg/l with TSAT < 20%) and presence of incomplete reverse remodeling (LVEF < 40%).
2. Age ≥18 years
3. Obtained informed consent
4. Stable pharmacological therapy of heart failure during the last 4 weeks (with the exception of diuretics)

Exclusion Criteria:

1. Hemochromatosis, iron overload, defined as TSAT > 45%
2. Hemoglobin > 15 g/dl at inclusion
3. Known hypersensitivity to injectafer®.
4. Known active infection, CRP>20 mg/L, clinically significant bleeding, active malignancy.
5. Chronic liver disease and/or screening alanine transaminase (ALT) or aspartate transaminase (AST) above three times the upper limit of the normal range.
6. Immunosuppressive therapy or renal dialysis (current or planned within the next 6 months).
7. History of erythropoietin, i. v. or oral iron therapy, and blood transfusion in previous 12 weeks and/or such therapy planned within the next 6 months.
8. Unstable angina pectoris as judged by the investigator, clinically significant uncorrected valvular disease or left ventricular outflow obstruction, obstructive cardiomyopathy, poorly controlled fast atrial fibrillation or flutter, poorly controlled symptomatic brady- or tachyarrhythmias.
9. Acute myocardial infarction or acute coronary syndrome, transient ischemic attack or stroke within the last 3 months.
10. Coronary-artery bypass graft, percutaneous intervention (e.g. cardiac, cerebrovascular, aortic; diagnostic catheters are allowed) or major surgery, including thoracic and cardiac surgery, within the last 3 months.
11. Inability to fully comprehend and/or perform study procedures in the investigator's opinion.
12. Vitamin B12 and/or serum folate deficiency according to the laboratory (re-screening is possible after substitution therapy).
13. Pregnancy or lactation.
14. Participation in another clinical trial within previous 30 days and/or anticipated participation in another trial during this study.
15. Planned cardiac hospitalization during study follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction from baseline | 3 months
  delta_LVEF measured by 3D-echocardiography

SECONDARY OUTCOMES:
Change in left ventricular end systolic volume from baseline | 3 months
  delta_LVESV measured by 3D-echocardiography
Change in left ventricular end diastolic volume from baseline | 3 months
  delta_LVEDV measured by 3D-echocardiography
Force frequency relationship | 3 months
  measured by 2D-echocardiography
Heart failure hospitalization and all-cause mortality | Up to six months
  measured by telephone contact
Incidence of Treatment-associated Serious and non-serious adverse events. | During intravenous study drug administration and 1-hour in hospital follow-up
  Serious and non-serious adverse events (AE) will be registered, which include:start date AE, duration AE, end-date AE, treatment group, continuation of AE after dose interruption, causality with study medication, presence of risk factors for AE and response to AE (sequela or recovery).

OTHER OUTCOMES:
Predefined right ventricular (RV) analysis | 3 months
  Assessment of effect of FCM on RV-function at rest and during incremental pacing. Assessment of RV-to-pulmonary artery coupling

CONTACTS AND LOCATIONS:
Locations (1):
- Pieter Martens, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Yes, full patient level data

REFERENCES:
- [Result] Martens P, Dupont M, Dauw J, Nijst P, Herbots L, Dendale P, Vandervoort P, Bruckers L, Tang WHW, Mullens W. The effect of intravenous ferric carboxymaltose on cardiac reverse remodelling following cardiac resynchronization therapy-the IRON-CRT trial. Eur Heart J. 2021 Dec 21;42(48):4905-4914. doi: 10.1093/eurheartj/ehab411. PMID 34185066